CLINICAL TRIAL: NCT03997799
Title: Comparison of Two Techniques of Video Assisted Thoracic Surgery (VATS) Uniportal Lobectomies Through the Transcervical and Standard Intercostal Approaches for Clinical Stage I Non-Small Cell Lung Cancer (NSCLC) in the Prospective Randomized Single-institutional Trial
Brief Title: Comparison of Two Techniques of Uniportal VATS Lobectomies for Clinical Stage I Non-Small Cell Lung Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pulmonary Hospital Zakopane (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 01/2019
Record Dates: First submitted 2019-06-18; First posted 2019-06-25 (Actual); Last update posted 2022-04-26 (Actual); Status verified 2022-04

CONDITIONS: Video Assisted Thoracic Surgery (VATS); Non-Small Cell Lung Cancer (NSCLC)
Keywords: lung cancer; mediastinum; pulmonary resection
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- uniportal transcervical approache (Experimental): Uniportal lobectomy with complete lymphadenectomy - transcervical approach with elevation of the sternum
  Interventions: Procedure: uniportal lobectomy with complete lymphadenectomy
- uniportal intercostal approache (Experimental): Uniportal lobectomy with complete lymphadenectomy - intercostal approache
  Interventions: Procedure: uniportal lobectomy with complete lymphadenectomy

INTERVENTIONS:
Procedure: uniportal lobectomy with complete lymphadenectomy — uniportal lobectomy with complete lymphadenectomy

SUMMARY:
Aim of the study is to compare safety and tolerance of two techniques of Video Assisted Thoracic Surgery (VATS) uniportal lobectomies in the prospective randomized single-institutional trial. One arm is a uniportal lobectomy performed through the transcervical approach with elevation of the sternum, the other arm will utilize a standard uniportal intercostal approache. There will be 10 patients in each group. Patients in clinical stage cI-III (T1-3N0-2M0) Non-Small Cell Lung Cancer (NSCLC). The results will be compared for time of the procedure, number of conversions to multi-portal VATS and/or open thoracotomy, duration and volume of chest drainage, amount of postoperatve pain, time of hospitalization and the number of resected lymph nodes and metastatic nodes. Accrual of patients is planned to complete within 12 months.

DETAILED DESCRIPTION:
Introduction Video-assisted thoracoscopic surgery (VATS) pulmonary lobectomy became an accepted method for the treatment of early-stage Non-Small-Cell Lung Cancer (NSCLC). There are several variants of VATS lobectomy. In recent years the uniportal approach described by Gonzales-Rivas gained a world-wide interest. The uniportal VATS approach can be performed through the intercostal incision as has been practiced in vast majority of published cases, but there is also another approach, namely the transcervical one, first described by Zakopane team in 2007. In that time, right upper lobectomy and afterwards the left upper lobectomy through the transcervical approach combined with single-port intercostal VATS were performed. The method was to combine lobectomy with Transcervical Extended Mediastinal Lymphadenectomy (TEMLA), preceding a pulmonary resection with intraoperative examination of the mediastinal nodes with the imprint cytology technique. From 2016, after adopting the technique of uniportal intercostal lobectomy, transcervical VATS uniportal lobectomies, without additional intercostal ports were performed. Now, resection of any rightsided or left-sided lobe with the transcervical approach are feasible to be performed.

Surgical Technique Preparation The patient is positioned supine on the operating table with a roll placed beneath the thoracic spine to elevate the chest and to hyperextend the patient's neck. Under general anaesthesia an endobronchial tube is inserted to conduct selective lung ventilation during the latter part of the procedure.

A transverse 6-8 cm transcervical collar incision is made in the neck in a standard way with division and suture-ligation of the anterior jugular veins bilaterally. The sternal manubrium is elevated with sharp one-tooth hook connected to the Zakopane II frame (Aesculap-Chifa, BBraun, Nowy Tomysl, Poland) to widen the access to the mediastinum. The first part of the procedure is TEMLA. The technique of this procedure, and possible pitfalls and the methods of management of intraoperative complications were published elsewhere [6]. In brief, the technique of TEMLA included dissection of all mediastinal nodal stations except for the pulmonary ligaments nodes (station 9). The subcarinal nodes, the periesophageal nodes, the right and left lower paratracheal nodes, and the right hilar nodes (stations 7, 8, 4R, 4L and 10R) were removed in the mediastinoscopy-assisted technique and the paraaortic and the pulmonary-window nodes (stations 6 and 5) are removed in the videothoracoscopy-assisted technique, with the videothoracoscope inserted through the transcervical incision. The superior mediastnal nodes and upper right and left paratracheal nodes (stations 1, 2R and 2L) are removed in the open surgery fashion under direct eye control. The prevascular and retrotracheal nodes (stations 3A and 3P) are removed in pre-selective cases. Generally, the mediastinal pleura is not violated and no drain is left in the mediastinum. Bilateral supraclavicular lymphadenectomy and even deep cervical lymph node dissection is possible during TEMLA through the same incision.

The nodes removed during TEMLA are sent sequentially to intraoperative pathologic examination with use of the imprint cytology technique [4]. The imprint cytology technique is a highly reliable technique much less time consuming than a frozen section analysis. Due to this advantage the time of nodal examinations adds only 15 to 20 minutes to the total time of the operation. After receiving the negative results of the imprint cytology, confirming there are no nodal metastasis the VATS lobectomy part starts. The position of the patient is slightly changed with the introduction of the roll beneath the patient's operating side. Additionally, the operating table is rotated to achieve a semi-lateral position of the patient. The ventillation of the operated lung is disconnected and the mediastinal pleura is opened. Further dissection is performed with the use of endostaplers to manage the lobar vesselts, bronchus and interlobar fissures.

ELIGIBILITY:
Inclusion Criteria:

- Patients with histologically, or cytologically proven clinical stage I (cI) NSCLC

Exclusion Criteria:

* Patients with more advanced NSCLC than clinical stage I (cI) NSCLC
* Severe atherosclerotic lesions of the innominate artery and the aortic arch and previous cardiac surgery.
* Severe pleural adhesions and calcified intrapulmonary nodes after previous tuberculosis are also technical obstacles for this kind of surgery.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-06-10 (Actual); Primary Completion 2019-06-10 (Actual); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
time of the procedure | 4 weeks
  duration of the operation in minutes
number of conversions to multi-portal VATS and/or open thoracotomy | 4 weeks
  number of conversions to multi-portal VATS and/or open thoracotomy
duration of chest drainage | 4 weeks
  duration of chest drainage in days
volume of chest drainage | 4 weeks
  volume of chest drainage in ml
amount of postoperatve pain | up to 72 hours after the end of surgery
  1.pain intensity 0-100 mm VAS scale measured every 4 hours on standard ruler beginning from the end of the surgery.
  The visual analogue scale (VAS) is commonly used as the outcome measure for such studies. It is usually presented as a 100-mm horizontal line on which the patient's pain intensity is represented by a point between the extremes of "no pain at all" and "worst pain imaginable." Its simplicity, reliability, and validity, as well as its ratio scale properties, make the VAS the optimal tool for describing pain severity or intensity.
time of hospitalization | 4 weeks
  time of hospitalization in days
number of resected lymph nodes | 4 weeks
  number of resected lymph nodes
number of resected metastatic nodes | 4 weeks
  number of resected metastatic nodes

CONTACTS AND LOCATIONS:
Overall Officials: Marcin Zielinski, MD PhD, Study Director — Pulmonary Hospital Zakopane
Locations (1):
- Pulmonary Hospital, Zakopane, Poland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Gonzalez D, Paradela M, Garcia J et al. Single-port video-assisted thoracoscopic lobectomy. Interact Cardiovasc Thorac Surg 2011;12:14-5 — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC3771611/
- See also: Zieliński M, Pankowski J, Hauer L et al: The right upper lobe pulmonary resection performed through the transcervical approach. Eur J Cardiothorac Surg. 2007;32:766-769 — https://www.ncbi.nlm.nih.gov/pubmed/17766130
- See also: Zieliński M, Nabialek T, Pankowski J. Transcervical uniportal pulmonary lobectomy. JOVS pulmonary transcervical J Vis Surg. 2018;4:42 — http://jovs.amegroups.com/article/view/18531/18723